CLINICAL TRIAL: NCT04762641
Title: A Phase 1 Dose Escalation and Expansion Study of ABL503, a Bispecific Antibody of 4-1BB and PD-L1, As a Single Agent in Subjects with Any Progressive Locally Advanced (unresectable) or Metastatic Solid Tumors
Brief Title: This is a Study to Evaluate the Safety and Tolerability of ABL503, and to Determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of ABL503 in Subjects with Any Progressive Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABL503-1001
Record Dates: First submitted 2021-01-28; First posted 2021-02-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABL503 (Experimental): ABL503 will be administered biweekly of every 28-day cycle in the dose-escalation. The dosing interval to be used in the dose-expansion part will be re-evaluated based on the emerging safety and PK data from the dose-escalation part of the study.
  Interventions: Drug: ABL503

INTERVENTIONS:
Drug: ABL503 — ABL503 will be administered intravenously (IV) on Day 1 and Day 15 of every 28-day cycle in the dose-escalation part. The dosing interval to be used in the dose-expansion part will be re-evaluated based on the emerging safety and PK data from the dose-escalation part of the study.

SUMMARY:
This is a first-in-human Phase 1, single-arm, open-label, multicenter, multiple-dose, dose-escalation and dose-expansion study of ABL503 to evaluate the safety, tolerability, MTD and/or RP2D, PK, immunogenicity, preliminary antitumor activity, and the PD effect of ABL503 in subjects with any progressive locally advanced (unresectable) or metastatic solid tumors who are relapsed or refractory following the last line of treatment and have no available standard of care option. This study includes 3 parts: a dose-escalation part, a dose-expansion part and tumor-expansion part

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed diagnosis of any progressive locally advanced (unresectable) or metastatic solid tumors that have relapsed or are refractory following the last line of treatment, for which prior standard therapy has been ineffective, standard therapy does not exist, or is not considered appropriate.
* With AE(s) excluding alopecia or Grade 2 toxicities that are deemed stable or irreversible (eg, peripheral neuropathy) from prior therapy that have improved to Grade 1 or the baseline grade more than 14 days prior to the first administration of the study drug
* Adequate hematologic, hepatic, and renal functions confirmed based on the screening laboratory tests and reconfirmed with additional safety laboratory tests performed within 72 hours prior to the first administration of ABL503

Exclusion Criteria:

* Prior anticancer monoclonal antibody treatment or investigational therapy within 28 days prior to the first administration of study drug or has not recovered (ie, ≤ Grade 1 or at baseline grade) from AEs due to previously administered agent more than 14 days prior to ABL503 administration
* Prior chemotherapy or radiation therapy within 2 weeks or targeted small molecule therapy within 5 half-lives prior to the first administration of study drug or has not recovered (ie, ≤ Grade 1 or at baseline grade) from AEs due to previously administered agent more than 14 days prior to ABL503 administration
* Requiring or received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration.
* Risk factors for bowel obstruction or bowel perforation (including but not limited to a history of acute diverticulitis, intra-abdominal abscess, and abdominal carcinomatosis.
* Discontinued from prior immunomodulatory therapy due to any intolerable immune-related adverse events (IrAEs) requiring systemic steroid treatment
* History of drug-induced pneumonitis (interstitial lung disease) or currently has pneumonitis
* Received prior treatment with an anti-4-1BB antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Dose-Limiting Toxicities (DLT) | From Day 1 until disease progression or Day 28, whichever came first
  Number of subjects with Dose-Limiting Toxicity (DLT)
Number of subjects with AE, IrAEs, IRRs, SAEs and abnormalities in Lab | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable AEs, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first, assessed up to approx. 12 months
  Number of subjects with Adverse Event, Immune-related Adverse Event, Infusion-related Reactions (IRRs), serious AEs, and abnormalities in lab parameters

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable AEs, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first, assessed up to approx. 12 months
  Proportion of subject with best overall response of complete response (CR) or partial response (PR) per RECIST v1.1
Pharmacokinetic (PK) of ABL503 | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable AEs, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first, assessed up to approx. 12 months
  Serum concentrations of ABL503 will be collected and analyzed to evaluate the PK of ABL503
Immunogenicity of ABL503 | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable AEs, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first, assessed up to approx. 12 months
  Incidence of anti-ABL503 antibody will be analyzed to evaluate the Immunogenicity of ABL503

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - City of Hope, Duarte, California
  - USC, Los Angeles, California
  - UCLA, Santa Monica, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - NEXT Oncology, San Antonio, Texas
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No